CLINICAL TRIAL: NCT06521086
Title: Optimizing Recovery in Trauma Patients: Integrating Enhanced Nutrition Delivery With Muscle Assessments, Functional Outcomes and Quality of Life
Brief Title: Optimizing Recovery in Trauma Patients by Integrating Enhanced Nutrition Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00114950
Record Dates: First submitted 2024-05-03; First posted 2024-07-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Trauma; Critical Illness
MeSH Terms: conditions — Wounds and Injuries; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Protein Supplementation (Experimental): Oral nutrition supplements (ONS) will be given, at maximum, three times per day throughout hospitalization. Upon discharge, participants will be given 4-weeks' worth of oral supplements to take. Adjustments may be made based on indirect calorimetry (IC) measurements.
  Interventions: Dietary Supplement: Nutrition Supplements - Fresubin KCAL Drinks
- Control Pathway (No Intervention): Standard of care nutrition delivery throughout hospitalization. Upon discharge participants will be sent home with standard nutrition information without Indirect Calorimetry (IC) guidance.

INTERVENTIONS:
Dietary Supplement: Nutrition Supplements - Fresubin KCAL Drinks — Fresubin drinks will be taken up to 3 times a day throughout hospitalization and for 4 weeks after discharge.
  Arms: Enhanced Protein Supplementation

SUMMARY:
This is a prospective, randomized, controlled trial designed to evaluate the impact of enhanced protein supplementation compared to a standard of care nutrition delivery in critically ill older adult trauma patients. Subjects will be randomized 1:1 to either enhanced nutrition or control arm. Subjects randomized to the enhanced nutrition arm will receive oral nutrition supplements (ONS) up to 3 times per day while in the hospital and for 4 weeks after discharge. Subjects in the standard of care arm will receive normal nutrition recommendations from their clinical providers. Participants in both groups will undergo non-invasive tests that measure how much energy (calories) they are using, body composition, and muscle mass.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled trial designed to evaluate the impact of enhanced protein supplementation compared to a standard of care nutrition delivery in critically ill older adult trauma patients. Enhanced protein supplementation supports patients from ICU admission to 4-weeks post-hospital discharge, providing a comprehensive and personalized plan of care carried to completion.

Subjects will be randomized 1:1 to enhanced nutrition or control arm. Subjects randomized enhanced nutrition oral nutrition supplements (Fresenius KCAL shakes) up to 3 times per day while in the hospital and for 4 weeks after discharge. Subjects in the standard of care arm will receive normal nutrition recommendations from their clinical providers.

Participants in both groups will undergo non-invasive tests that measure how much energy (calories) they are using, body composition, and muscle mass. They will also be asked to complete walking and strength tests, and surveys about quality of life.These will be done at hospital admission, day 14 or hospital discharge, and at a one month post-discharge follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 45 years old and presented to the Emergency Department as a leveled trauma
* Patients who have the ability to tolerate oral nutrition
* Patients who have had a standard of care CT scan this admission

Exclusion Criteria:

* Expected withdrawal of life-sustaining treatment within 48 hours
* Traumatic Brain Injury
* Presence of lower extremity fracture(s)
* Mechanical Ventilation
* Subjects for who the Investigator would recommend a different supplement based on their medical condition.
* Prisoner
* Pregnancy for women of child-bearing potential

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in muscle mass as a measure of muscle quality | Baseline to one month post-discharge (approximately six weeks)
Change in glycogen stores as a measure of muscle quality | Baseline to one month post-discharge (approximately six weeks)
Change in body composition (percentage of a body's weight that is fat tissue) as a measure of muscle quality | Baseline to one month post-discharge (approximately six weeks)
  Body composition is the percentage of a body's weight that is fat tissue.

SECONDARY OUTCOMES:
Change in six minute walk test (6MWT) distance | Baseline to one month post-discharge (approximately six weeks)
  The 6MWT assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.
Change in four meter gait speed | Baseline to one month post-discharge (approximately six weeks)
  Four meter gait speed is the time one takes to walk four meters on a level surface.
Change in 30-second sit to stand test | Baseline to one month post-discharge (approximately six weeks)
  This test measures the number of times an individual can stand from a chair with no assistance in 30 seconds. This test is used to assess functional lower body strength.
Change in grip strength | Baseline to one month post-discharge (approximately six weeks)
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength.
Change in quadriceps strength | Baseline to one month post-discharge (approximately six weeks)
  ED (electromechanical dynamometry) can be used in either isometric or isokinetic mode. Quadriceps strength is expressed as peak knee extensor torque, which is produced at around 60° knee flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No